CLINICAL TRIAL: NCT05807698
Title: The Effect of Laughter Yoga on Psychological Well-Being and Quality of Life in Physically Disabled Women and Their Relatives
Brief Title: The Effect of Laughter Yoga on Psychological Well-Being
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinop University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: sinopUberna-2
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Laughter; Quality of Life
Keywords: laughter therapy; psychological well being; quality of life; Physically Disabled Women
MeSH Terms: conditions — Laughter; Psychological Well-Being | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): Assigned Interventions Laughter therapy session will be applied online for 25-30 minutes once a week for 2 months by the researcher who has the Laughter therapy certificate to the application group. In the laughter therapy session, the practices of introducing the practitioner and introducing the therapy, breathing exercises for a healthy life, keeping the rhythm accompanied by music, turning the laughter that started as if it were childlike games into reality will be carried out.
  Interventions: Behavioral: laughter therapy

INTERVENTIONS:
Behavioral: laughter therapy — Assigned Interventions Laughter therapy session will be applied online for 25-30 minutes once a week for 2 months by the researcher who has the Laughter therapy certificate to the application group. In the laughter therapy session, the practices of introducing the practitioner and introducing the therapy, breathing exercises for a healthy life, keeping the rhythm accompanied by music, turning the laughter that started as if it were childlike games into reality will be carried out.

SUMMARY:
Brief Summary: The definition of individuals with disabilities, who are among the disadvantaged group, is defined by Law No. 5378 as "those who have difficulties in adapting to social life and meeting their daily needs due to the loss of their physical, mental, spiritual, sensory and social abilities at various degrees due to any congenital or subsequent reason; and a person who needs protection, care, rehabilitation, counseling and support services" (Law on the Disabled).

Due to the fact that the conditions and needs of physically disabled women are not well expressed, they have not benefited enough from services such as education and health and they have faced difficulties. No study has been found in the world or in our country that examines the effect of laughter yoga on physically disabled women and their relatives. In this study, it is thought that the practice of laughter yoga can increase the psychological well-being and quality of life of physically disabled women and their relatives.

Aim: This study was planned to measure the effect of laughter yoga on psychological well-being and quality of life in physically disabled women and their relatives.

DETAILED DESCRIPTION:
Detailed Description: Method: The research was planned as a quasi-experimental study including pre-test, post-test and follow-up.

The research will be carried out by reaching physically disabled women and their relatives affiliated to Sinop Disabled Association.

Population and Sample: Disabled women living and their relatives in Sinop in the Sinop Disabled Association will form the universe of our study, and all individuals who have agreed to participate in the study and volunteered will form the sample.

How the research was conducted: Laughter yoga to be done will last eight weeks, once a week. Each session of laughter yoga is planned to be approximately 40 minutes. Personal Information Form, Psychological Well-Being Scale, SF-12 Quality of Life Scale Short Form, Psychological Well-Being Scale and SF-12 Quality of Life Scale as a post-test at the end of the laughter yoga were used for the physically disabled women and their relatives who agreed to participate in the study before starting the study. The Short Form and the Psychological Well-Being Scale and the SF-12 Quality of Life Scale Short Form will be administered again in the follow-up (one month after the application has ended).

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Being woman,
* Not being mentally handicapped
* Having a physical disability
* Being a relative caring for a woman with a physical disability.

Exclusion Criteria:

* Not being between the ages of 18-65,
* To being male,
* Being mentally handicapped
* Not having a physical disability
* Not volunteering to participate in the research.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-10 (Estimated); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Psychological Well-Being Scale | one day
  It was developed by Diener et al., (2010) and adapted into Turkish by Telef (2013). It is a single factor, 7-point Likert scale consisting of 8 items. The range of scores obtained varies between 8 and 56. A high score from the scale indicates that the individual is psychologically strong.

SECONDARY OUTCOMES:
SF-12 Quality of Life Scale Short Form | one day
  The scale includes physical functioning (questions 2a, 2b, 2 and 3), physical role (questions 2, 3a, 3b, 4 and 5), body pain (1 item 5, 8th question), general health (1 item 1, 1st question), energy (1 item 6b, 10th question), social functionality (1 item, 7, 12th question), emotional role (2 items 4a 4b, 6 and 7th question) and mental health (2 items 6a, 6c, 9 and 11 items) and 8 sub-dimensions and 12 items. Items related to physical and emotional role were answered as dichotomy (yes or no), while other items had Likert type options ranging between 3 and 6. While the FIM-12 score is obtained from the sub-dimensions of general health, physical functionality, physical role and body pain, the MBS-12 score is obtained from the sub-dimensions of social functionality, emotional role, mental health and energy. Both FIM-12 and DRD-12 scores range from 0 to 100, with higher scores representing better health.

CONTACTS AND LOCATIONS:
Overall Officials: Berna ERSOY ÖZCAN, PhD, Principal Investigator — Sinop University; Yasemin ÖZYER, PhD, Principal Investigator — Sinop University

IPD SHARING:
Plan to Share IPD: No